CLINICAL TRIAL: NCT00815672
Title: The Influence of Home-based Aerobic and Resistance Exercise on Cancer-Related Fatigue, Strength, and Muscle Mass in Prostate Patients.
Brief Title: Exercise for Prostate Cancer Patients
Acronym: EXCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Karen Mustian, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1703DOD
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2018-11

CONDITIONS: Fatigue
Keywords: Exercise; Prostate cancer; Fatigue
MeSH Terms: conditions — Fatigue; Motor Activity; Prostatic Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Arm 1 (No Intervention): Usual Care: Standard care monitoring
- Treatment arm 2 (Experimental): Home-based Exercise: Progressive walking and resistance exercise treatment.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Progressive walking and resistance exercise treatment
  Arms: Treatment arm 2

SUMMARY:
The purpose of this study is to gain a better understanding of the mechanisms responsible for cancer-related fatigue.

DETAILED DESCRIPTION:
Numerous studies have shown that the vast majority of patients experience cancer-related fatigue (CRF) during cancer treatments. Research by our group showed that 71% percent of 84 prostate cancer patients reported CRF during radiation. Unlike fatigue caused by overexertion, CRF is a pervasive, whole-body experience that is not alleviated by rest or sleep and often lingers long after completing standard treatments like radiation therapy. It has a detrimental effect on patients' quality of life and can interfere with completion of prescribed treatment regimens. In addition, lasting fatigue for many patients impedes the resumption of normal life following treatments. Unfortunately, effective, well-accepted treatments for CRF are lacking. Although some research suggests that exercise may be a promising intervention for reducing CRF, physicians are still hesitant to prescribe exercise for fatigued patients, and, in fact, often encourage them to rest and conserve energy, which may be in exact opposition to what is needed.

One probable peripheral physiological mechanism that may affect the influence CRF is a loss of skeletal muscle mass, which, ultimately, effects weakness and strength. This muscle loss can result from deconditioning effects stemming from reduced physical activity resulting from cancer and its treatment. It is plausible that patients may enter radiation therapy with a certain degree of muscle loss, reduced strength and substantially decreased levels of physical activity as a result of their cancer diagnosis and the associated stress, surgical and systemic treatments, and/or the subsequent symptomology. Additionally, their physical activity may decline even further during radiation and escalate the loss of muscle and decreased strength. Recently, researchers have proposed that these deconditioning responses, as well as generalized inflammatory responses resulting from the cancer and/or its treatment result in skeletal muscle loss and strength deficits, which may play a significant role in the etiology of CRF. Although mild exercise can counteract deconditioning, current research has shown that cancer patients decrease the amount of physical activity they engage in after diagnosis as well as during and after treatment. Additionally, a substantial number of patients never return to prediagnosis levels of physical exercise and do not meet the minimal ACSM or CDC guidelines for achieving the health-related benefits (e.g., increased muscle mass, strength, and cardiorespiratory fitness) thought to be etiologically involved in CRF, suggesting the need for formal intervention.

We propose to test an individually tailored physical exercise intervention, including both aerobic and resistance exercise, for reducing CRF in prostate cancer patients receiving radiation therapy. The proposed research will provide detailed information on the efficacy and acceptance of a home-based aerobic and resistance exercise program for CRF among prostate cancer patients receiving radiation. Data regarding the influence of this intervention on potential factors related to CRF, including loss of strength, muscle atrophy and inflammatory biomarkers will be gathered. The purpose of the proposed study is to extend the positive findings from a feasibility study showing that our tailored home-based aerobic (walking) and progressive resistance exercise program was effective in reducing CRF and improving strength, skeletal muscle mass, aerobic capacity and quality of life in a small sample of prostate and breast cancer patients (N=38).

The Primary Aim of the study is to examine the influence of a home-based aerobic and progressive resistance exercise program on CRF in prostate cancer patients receiving radiation therapy. The proposed study is a phase II randomized, 2-arm, controlled clinical trial employing a repeated-measures design (baseline, post intervention, 3-month follow-up) that will accrue 122 male prostate cancer patients receiving radiation therapy.

This project builds upon very promising pilot data and includes a diverse research team with substantial experience in exercise interventions, survivorship, and cancer control research. This grant will allow us to discern the efficacy of a novel, tailored, home-based aerobic and resistance exercise intervention for reducing CRF among prostate cancer patients during radiation, and to identify potential factors (e.g., loss of strength, muscle atrophy, dysregulation of bodily immune function} that may contribute to the development of CRF that, in turn, can be more effectively targeted through tailoring future exercise interventions to improve the impact of these exercise interventions on reducing CRF. These results will have the direct potential to reduce the suffering experienced by prostate cancer patients during radiation treatments, and to positively impact future research in exercise and cancer control on side effect management, the practice of evidence-based medicine for the treatment of CRF, and, eventually, public health policy and oncology practice.

ELIGIBILITY:
Inclusion Criteria:

* Have a primary diagnosis of prostate cancer
* Have a KPS of 60 or greater.
* Be receiving any form of treatment for their prostate cancer or have received some form of treatment (e.g. surgery, chemotherapy, radiation therapy, hormone therapy) in the last 10 years
* Have approval of physician and be able to read English.
* Be 21 years of age or older and give informed consent

Exclusion Criteria:

* Have bone metastases that preclude participation due to symptoms such as pain or location of the bone metastasis.
* Have physical limitations that contraindicate participation.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-12; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Cancer-related fatigue | 4.5 Months
  The primary outcome measure for this study is CRF assessed by the FACIT-F fatigue subscale at the end of the 6th calendar week of the study.

SECONDARY OUTCOMES:
To provide preliminary data on influence of home-based aerobic and resistance exercise on the following: Strength | 4.5 months
  Strength: 7-10 repetition maximum test
To provide preliminary data on influence of home-based aerobic and resistance exercise on the following: Skeletal Muscle Mass | 4.5 months
  Skeletal Muscle Mass: DEXA
To provide preliminary data on influence of home-based aerobic and resistance exercise on the following: QOL | 4.5 months
  QOL: Facit-F
To provide preliminary data on influence of home-based aerobic and resistance exercise on the following: Sleep Quality | 4.5 months
  Sleep Quality: PSQI
To provide preliminary data on influence of home-based aerobic and resistance exercise on the following: Self Esteem | 4.5 months
  Self Esteem: RSE
To provide preliminary data on influence of home-based aerobic and resistance exercise on the following: Inflammatory Cytokines | 4.5 months
  Inflammatory Cytokines: Cytokine Specific ELISAs

CONTACTS AND LOCATIONS:
Overall Officials: Karen Mustian, Ph.D., Principal Investigator — James P. Wilmot Cancer Center, University of Rochester
Locations (1):
- James P. Wilmot Cancer Center, University of Rochester, Rochester, New York, United States